CLINICAL TRIAL: NCT00781196
Title: Effect of Low Dose Oral Folic Acid Supplementation on Phenytoin Induced Gingival Overgrowth: A Randomized Double Blind Controlled Trial.
Brief Title: Folic Acid Supplementation in Phenytoin Induced Gingival Overgrowth
Acronym: PIGO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Ravindra Arya, All India Institute of Medical Sciences, New Delhi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PIGO
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Gingival Overgrowth
Keywords: phenytoin; gum hyperplasia; phenytoin induced gingival overgrowth; plaque index; gingival overgrowth grade
MeSH Terms: conditions — Gingival Overgrowth; Gingival Hyperplasia | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Oral folic acid
  Interventions: Drug: folic acid
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: folic acid — capsule 0.5 mg once a day
  Arms: 1
Drug: placebo — capsule, once a day
  Arms: 2

SUMMARY:
Phenytoin, a common anti-seizure drug, leads to cosmetically unacceptable side effect of gingival overgrowth in a significant number of patients. There is some evidence of therapeutic effect of folic acid in cases of established phenytoin induced gingival overgrowth. In this study, the aim is to study the prospective preventive effect of low dose oral folic acid supplementation on phenytoin induced gingival overgrowth in epileptic children.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-15 yr
* Started on phenytoin within 1 mo of enrollment

Exclusion Criteria:

* Not willing to participate
* On other folic acid antagonists e.g. anti-neoplastic drugs for >/= 2 wks during last 3 months
* Pre-existing gingival over-growth due to other cause

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of any grade of overgrowth in 2 groups after 6 mo of phenytoin therapy | 6 months

SECONDARY OUTCOMES:
Occurrence of grade > 2 hyperplasia at the end of 6 mo | 6 months
Time to occurrence of grade > 2 overgrowth | open
Correlation between following and occurrence of grade > 2 overgrowth *phenytoin dose (in mg/kg/d) *serum phenytoin levels *plaque index | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Arya R, Gulati S, Kabra M, Sahu JK, Kalra V. Folic acid supplementation prevents phenytoin-induced gingival overgrowth in children. Neurology. 2011 Apr 12;76(15):1338-43. doi: 10.1212/WNL.0b013e3182152844. PMID 21482950